CLINICAL TRIAL: NCT04718311
Title: Analysis of Two Treatment Protocols for Patients With Oral Lichen Planus
Brief Title: Study on Treatment for Patients With Symptomatic Oral Lichen Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Researcher, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 121/120
Record Dates: First submitted 2021-01-16; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Lichen Planus, Oral
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tacrolimus treatment (Active Comparator): Apply a small amount (about 1 teaspoon) of medication to the lesions, twice a day after brushing the teeth, with a soft bristle toothbrush or with a finger (covered with a well-fitting glove).
  Interventions: Drug: Oral lichen clinical Healing evaluation
- Anti-inflammatory mouthwash (Placebo Comparator): Anti-inflammatory mouthwash In patients of the anti-inflammatory group, the mouthwash was used pure and without dilution at a dosage of 20 ml 3 times a day, immediately after normal daily oral hygiene was prescribed. It contains calcium hydroxide, hyaluronic acid, Umbelliferone and Oligomeric Proanthocyanidins. Patients were instructed to rinse for at least 5 minutes over the entire oral mucosa, with particular emphasis on the regions where the lesions are located.
  Interventions: Drug: Oral lichen clinical Healing evaluation

INTERVENTIONS:
Drug: Oral lichen clinical Healing evaluation — Treatments were topically applied for 5 days
  Other Names: Topical drug tacrolimus or mouthwash application

SUMMARY:
The primary objective of this study was to compare the therapeutic efficacy of Tacrolimus gel versus an anti-inflammatory mouthwash in an oral solution for the management of patients suffering from symptomatic OLP. The secondary objective was to analyze which one of the two treatments induced a greater risk of developing side effects.

DETAILED DESCRIPTION:
Thirty nine patients were assigned, through a randomized design, to receive tacrolimus ointment 0.1% or a mouthwash composed of calcium hydroxide 10%, hyaluronic acid 0,3%, umbelliferone and oligomeric proanthocyanidins, or an anti-inflammatory mouthwash (mouthwash which contains calcium hydroxide, hyaluronic acid, Umbelliferone and Oligomeric Proanthocyanidins) for 3-months. At baseline (T0) and after 3 months (T1), patients were subjected to clinical and oral assessments and were evaluated for the symptoms (Numerical Pain Scale, NRS score) and signs (Thongprasom's score) of OLP. Data were calculated using T-test for the dependent variable, Wilcoxon test and Mann-Witney u test.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* clinical diagnosis and histological diagnosis of OLP on the basis of WHO criteria;
* presence of symptoms related to OLP.

Exclusion Criteria:

* presence of systemic conditions that may have affected the study results;
* state of pregnancy or breastfeeding;
* histological signs of dysplasia;
* drugs inducing a lichen response (ACE-inhibitors, β-blockers, etc.);
* treatment of OLP in the six months prior to the start of the programme;
* presence of extraoral lesions (genital, skin and other)
* history of previous immunodeficiency or HIV seropositivity;
* previous allogeneic bone marrow transplantation;
* presence of systemic lupus erythematosus or other autoimmune diseases.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Clinical Mucosal healing | 180 days
  Patients clinically were evaluated using the scale used by Thongprasom et al. as reference. This gives a score that varies from 0 to 5, using a millimetre reference: 0, in the absence of lesions; 1, in the presence of hyperkeratosis streaks; 2, in the presence of an atrophic area less than 1 mm2; 3, in the presence of an atrophic area greater than
  1 mm2; 4, in the presence of an erosive area less than 1 mm2; 5, in the presence of an erosive area greater than 1 mm2. In the presence of multiple injuries, the value has been calculated by summing the values of each injury.

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — Università degli Studi di Catania
Locations (1):
- University of Catania, Catania, CT, Italy

IPD SHARING:
Plan to Share IPD: Yes
Sharing results
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: pubmed